CLINICAL TRIAL: NCT06000059
Title: Mental Health Stigma in Rural Uganda
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Empower Through Health (Unknown); Empowerment to Heal - Uganda (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000034605; No NIH funding (Other: 01.22.24)
Record Dates: First submitted 2023-08-10; First posted 2023-08-21 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Mental Health Issue

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Radio Drama (Experimental): Participants in this group will participate in three listening sessions. The first and third listening sessions will consist of information unrelated to mental illness. The second listening session will be the radio theater intervention that is being developed.
  Interventions: Behavioral: Radio Drama
- Control (No Intervention): Participants in this group will participate in three listening sessions all unrelated to mental illness.
- Randomly selected community members (No Intervention): randomly selected members of the community that have not had exposure to the intervention over the course

INTERVENTIONS:
Behavioral: Radio Drama — An hour long radio drama adapted from from a previous community-led theater intervention
  Arms: Radio Drama

SUMMARY:
The investigators aim to elucidate attitudes and stigma towards mental illness in the pathways to mental healthcare among key stakeholders, such as traditional healers, religious leaders, families of those with mental illness, and those with mental illness. Investigators also will measure the levels of stigma expressed by members of the general community based on gender of the individual with mental illness and the specific mental health condition. Additionally, the investigators hope to convert the previously conducted theater intervention to a radio production, which is the most commonly used form of media in Uganda, and test its effectiveness for changing attitudes and reducing stigma towards mental illness throughout society.

DETAILED DESCRIPTION:
The scientific objective of this protocol is to develop and evaluate a novel intervention to reduce mental illness stigma among people in rural Uganda. The central hypothesis to be assessed is that a community-designed radio-based intervention can decrease mental illness stigma and lead to improved health-seeking behaviors. This hypothesis is supported by preliminary data demonstrating for the first time, to our knowledge, the effectiveness of an arts intervention to reduce mental health stigma in the general population in a rural region of a low income country. The investigators drew on message design theory underpinned by an audience-channel-message-evaluation (ACME) framework to design the intervention, a community-led theater performance in collaboration with community health workers in the rural Busoga Region of Eastern Uganda.

Radio is also popular in Uganda, with 78% of all Ugandans in rural and urban areas alike report listening to the radio. Listening to the radio is often a social activity. Adapting the ACME framework, the investigator will work with the community to convert their previously tested theater intervention into a radio intervention that can be deployed at scale.

Additionally, to better target future anti-stigma interventions, investigators will measure how the levels of stigma endorsed by the general community differ based on the mental health condition and the gender of those with mental illness.

Aim 1: Develop a radio drama derived from our previous theater intervention designed to decrease community stigma towards mental illness and increase healthcare seeking behaviors among those with mental illness.

Aim 2: Utilize qualitative methods, such as focus groups and in-depth interviews, to explore local responses to the radio drama and aspects fostering its acceptance or rejection.

Aim 3: Use a cluster randomized control trial to test the effectiveness of the radio drama in decreasing mental illness stigma immediately post-intervention and at one-month follow-up.

Aim 4: Evaluate levels of stigma endorsed by general community based on mental health condition and the gender of those with mental illness.

Hypothesis: Participants randomized to the radio drama intervention will show lower levels of mental illness stigma, compared with the control group.

The focus of this registration is Aim 3.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be willing to fully participate in the study - for the radio stigma intervention, it will include three separate listening sessions and two structured questionnaires. For evaluation of differential levels of stigma based on gender and condition, it will include listening to vignettes portraying mental illness and answering a questionnaire
* All members must reside in the village where the intervention is being conducted.
* Individuals must be able to provide written informed consent.

Exclusion Criteria:

* Those who cannot or are not able to willingly give consent to participate in this study will be excluded.
* Individuals who already have a family member participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Broad Acceptance Scale (BAS) | baseline and 1 month post intervention, an average of 2 months
  The BAS is a 10-item questionnaire targeted to structural stigma, the "societal-level conditions, cultural norms, and institutional practices that constrain the opportunities, resources, and wellbeing" for individuals with mental illness. Each yes adds one point to the scale, and five questions from each scale were reverse-scored to match the direction of the scale. There were ten questions, therefore it generated a score between zero and ten. Higher scores indicated more acceptance and less stigma towards mental illness, while lower scores indicated less acceptance and more stigma towards mental illness.
Change in Personal Acceptance Scale (PAS) | baseline and 1 month post intervention, an average of 2 months
  The PAS is a 9-item questionnaire targeted to public stigma, the "negative attitudes, beliefs, and behaviors held within a community" against individuals with mental illness. Each yes adds one point to the scale, and five questions from each scale were reverse-scored to match the direction of the scale. The total number of points was divided by the number of questions (nine) and multiplied by ten to generate numbers between zero and ten for comparison purposes to the Broad Acceptance Scale. Higher scores indicated more acceptance and less stigma towards mental illness, while lower scores indicated less acceptance and more stigma towards mental illness.

SECONDARY OUTCOMES:
Change in Broad Acceptance Scale (BAS) | baseline and up to one year
  BAS will be calculated for randomly selected community members based on the mental health condition and the gender of those with mental illness. The BAS is a 10-item questionnaire targeted to structural stigma, the "societal-level conditions, cultural norms, and institutional practices that constrain the opportunities, resources, and wellbeing" for individuals with mental illness. Each yes adds one point to the scale, and five questions from each scale were reverse-scored to match the direction of the scale. There were ten questions, therefore it generated a score between zero and ten. Higher scores indicated more acceptance and less stigma towards mental illness, while lower scores indicated less acceptance and more stigma towards mental illness.
Change in Personal Acceptance Scale (PAS) | baseline and up to one year
  PAS will be calculated for randomly selected community members based on the mental health condition and the gender of those with mental illness. The PAS is a 9-item questionnaire targeted to public stigma, the "negative attitudes, beliefs, and behaviors held within a community" against individuals with mental illness. Each yes adds one point to the scale, and five questions from each scale were reverse-scored to match the direction of the scale. The total number of points was divided by the number of questions (nine) and multiplied by ten to generate numbers between zero and ten for comparison purposes to the Broad Acceptance Scale. Higher scores indicated more acceptance and less stigma towards mental illness, while lower scores indicated less acceptance and more stigma towards mental illness.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Jae Lee, MD, Principal Investigator — Yale University
Locations (1):
- Empowerment to Heal - Uganda, Mpunde, Buyende District, Uganda